CLINICAL TRIAL: NCT01787799
Title: EVOLVE II QCA: A Prospective, Multicenter Trial to Assess the SYNERGY Everolimus-Eluting Platinum Chromium Coronary Stent System (SYNERGY Stent System) for the Treatment of Atherosclerotic Lesion(s)
Brief Title: EVOLVE II QCA: A Prospective, Multicenter Trial to Assess the SYNERGY Stent System for the Treatment of Atherosclerotic Lesion(s)
Acronym: EVOLVE II QCA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: Beth Israel Deaconess Medical Center (Other); Medstar Health Research Institute (Other); Quintiles, Inc. (Industry); Medidata Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2072
Record Dates: First submitted 2013-01-16; First posted 2013-02-11 (Estimated); Results first posted 2016-03-16 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-02

CONDITIONS: Atherosclerotic Lesion(s)
Keywords: Drug-eluting stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SYNERGY Stent System (Experimental): SYNERGY Everolimus-Eluting Platinum Chromium Coronary Stent System (SYNERGY Stent System)
  Interventions: Device: SYNERGY

INTERVENTIONS:
Device: SYNERGY — Synergy is a device/drug combination product composed of two components, a device (coronary stent system including a chromium stent platform) and a drug product (a formulation of everolimus contained in a bioabsorbable polymer coating.

SUMMARY:
The purpose of this study is to evaluate 9 month angiographic and intravascular ultrasound (IVUS) data for the SYNERGY Everolimus-Eluting Platinum Chromium Coronary Stent System (SYNERGY Stent System) in the treatment of subjects with atherosclerotic lesion(s) ≤34 mm in length (by visual estimate) in native coronary arteries ≥2.25 mm to ≤4.0 mm in diameter (by visual estimate).

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years of age
* Subject (or legal guardian) understands the trial requirements and the treatment procedures and provides written informed consent before any trial-specific tests or procedures are performed
* For subjects less than 20 years of age enrolled at a Japanese site, the subject and the subject's legal representative must provide written informed consent before any study-specific tests or procedures are performed
* Subject is eligible for percutaneous coronary intervention (PCI)
* Subject has symptomatic coronary artery disease with objective evidence of ischemia or silent ischemia
* Subject is an acceptable candidate for coronary artery bypass grafting (CABG)
* Subject is willing to comply with all protocol-required follow-up evaluation

Angiographic Inclusion Criteria (visual estimate)

* Target lesion(s) must be located in a native coronary artery with a visually estimated reference vessel diameter (RVD) ≥2.25 mm and ≤4.0 mm
* Target lesion(s) length must be ≤34 mm (by visual estimate)
* Target lesion(s) must have visually estimated stenosis ≥50% and <100% with thrombolysis in Myocardial Infarction (TIMI) flow >1 and one of the following (stenosis ≥70%, abnormal fractional flow reserve (FFR), abnormal stress or imaging stress test, or elevated biomarkers prior to the procedure)
* Coronary anatomy is likely to allow delivery of a study device to the target lesions(s)
* The first lesion treated must be successfully pre-dilated/pretreated

Exclusion Criteria:

* Subject has clinical symptoms and/or electrocardiogram (ECG) changes consistent with acute ST elevation MI (STEMI)
* Subject has cardiogenic shock, hemodynamic instability requiring inotropic or mechanical circulatory support, intractable ventricular arrhythmias, or ongoing intractable angina
* Subject has received an organ transplant or is on a waiting list for an organ transplant
* Subject is receiving or scheduled to receive chemotherapy within 30 days before or after the index procedure
* Planned PCI (including staged procedures) or CABG after the index procedure
* Subject previously treated at any time with intravascular brachytherapy
* Subject has a known allergy to contrast (that cannot be adequately premedicated) and/or the trial stent system or protocol-required concomitant medications (e.g., platinum, platinum-chromium alloy, stainless steel, everolimus or structurally related compounds, polymer or individual components, all P2Y12 inhibitors (clopidogrel, ticlopidine, prasugrel, or ticagrelor), or aspirin)
* Subject has one of the following (as assessed prior to the index procedure):

  * Other serious medical illness (e.g., cancer, congestive heart failure) with estimated life expectancy of less than 24 months
  * Current problems with substance abuse (e.g., alcohol, cocaine, heroin, etc.)
  * Planned procedure that may cause non-compliance with the protocol or confound data interpretation
* Subject is receiving chronic (≥72 hours) anticoagulation therapy (i.e., heparin, coumadin) for indications other than acute coronary syndrome
* Subject has a platelet count <100,000 cells/mm3 or >700,000 cells/mm3
* Subject has a white blood cell (WBC) count < 3,000 cells/mm3
* Subject has documented or suspected liver disease, including laboratory evidence of hepatitis
* Subject is on dialysis or has baseline serum creatinine level >2.0 mg/dL (177µmol/L)
* Subject has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions
* Subject has had a history of cerebrovascular accident (CVA) or transient ischemic attack (TIA) within the past 6 months
* Subject has an active peptic ulcer or active gastrointestinal (GI) bleeding
* Subject has severe symptomatic heart failure (i.e., New York Heart Association (NYHA) class IV)
* Subject is participating in another investigational drug or device clinical trial that has not reached its primary endpoint
* Subject intends to participate in another investigational drug or device clinical trial within 12 months after the index procedure
* Subject with known intention to procreate within 12 months after the index procedure (women of child-bearing potential who are sexually active must agree to use a reliable method of contraception from the time of screening through 12 months after the index procedure)
* Subject is a woman who is pregnant or nursing (a pregnancy test must be performed within 7 days prior to the index procedure in women of child-bearing potential)

Angiographic Exclusion Criteria (visual estimate)

Planned treatment of more than 3 lesions

* Planned treatment of lesions in more than 2 major epicardial vessels
* Planned treatment of a single lesion with more than 1 stent
* Subject has 2 target lesions in the same vessel that are separated by less than 15 mm (by visual estimate)
* Target lesion(s) is located in the left main
* Target lesion(s) is located within 3 mm of the origin of the left anterior descending (LAD) coronary artery or left circumflex (LCx) coronary artery by visual estimate.
* Target lesion(s) is located within a saphenous vein graft or an arterial graft
* Target lesion(s) will be accessed via a saphenous vein graft or arterial graft
* Target lesion(s) with a TIMI flow 0 (total occlusion) or TIMI flow 1 prior to guide wire crossing
* Target lesion(s) treated during the index procedure that involves a complex bifurcation (e.g., bifurcation lesion requiring treatment with more than 1 stent)
* Target lesion(s) is restenotic from a previous stent implantation or study stent would overlap with a previous stent
* Subject has unprotected left main coronary artery disease (>50% diameter stenosis)
* Subject has been treated with any type of PCI (i.e., balloon angioplasty, stent, cutting balloon atherectomy) within 24 hours prior to the index procedure
* Thrombus, or possible thrombus, present in the target vessel (by visual estimate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-03; Primary Completion 2014-08 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Meredith, Professor, Principal Investigator — Monash Medical Centre-Clayton Campus, 246 Clayton Road, 3168 Clayton, Victoria, Australia
Locations (13):
- Australia (4):
  - The Prince Charles Hospital, Chermside, Queensland
  - Monash Medical Centre-Clayton Campus, Clayton, Victoria
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Fremantle Hospital, Fremantle, Western Australia
- Shonan Kamakura General Hospital, Kamakura-shi, Kanagawa, Japan
- New Zealand (6):
  - Mercy Angiography Unit, Ltd., Auckland
  - Auckland City Hospital, Auckland
  - Ascot Angiography Ltd, Auckland
  - Middlemore Hospital, Auckland
  - North Shore Hospital, Auckland
  - Christchurch Hospital NZ, Christchurch
- Singapore (2):
  - National University Hospital, Singapore
  - National Heart Centre, Singapore

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 100 subjects were enrolled at 12 centers in Australia, New Zealand, Singapore and Japan between March 25, 2013 and October 15, 2013.
Period: Overall Study
Arm/Group | SYNERGY Stent System
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Subjects greater than or equal to 18 years of age with symptomatic coronary artery disease with objective evidence of ischemia or silent ischemia. Subjects received the SYNERGY stent system for treatment of atherosclerotic lesion(s) less than or equal to 34mm in length and between 2.25mm and 4.0mm in diameter, both by visual estimate.
Arm/Group | SYNERGY Stent System
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.49 (10.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 80
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0
  Asian | 28
  Black, of African Heritage | 0
  Caucasian | 70
  Hispanic or Latino | 0
  Native Hawaiian or other Pacific Islader | 0
  Other | 2
  Not disclosed | 0
Region of Enrollment [Number; unit: participants]
  New Zealand | 69
  Singapore | 11
  Japan | 10
  Australia | 10
Cardiac Risk Factors [Number; unit: participants] — The same participant may be included in more than one category therefore the number of participants does not equal the total number of participants in the group.
  participants
    Hyperlipidemia Requiring Medication | 90
    Hypertension Requiring Medication | 71
    Family History of Coronary Artery Disease | 57
    History of PCI | 33
    History of Myocardial Infarction | 18
    Current Diabetes Mellitus; Medically Treated | 17
Lesion Characteristics [Mean (Standard Deviation); unit: mm]
  Reference Vessel Diameter | 2.66 (0.46)
  Lesion Length | 14.38 (7.49)
  Minimum Lumen Diameter | 0.86 (0.28)
  Percent Diameter Stenosis | 67.54 (9.59)

OUTCOME MEASURES:

1. Primary Outcome: In-stent Late Loss
Description: In-stent late loss at 9 months post-procedure as measured by quantitative coronary angiography (QCA)
Time Frame: 9 month
Population: The primary endpoint would be considered to have been met if the SYNERGY in-stent late loss was less than the performance goal of 0.40 mm. The Intent To Treat (ITT) and per protocol populations were identical.
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | SYNERGY Stent System
Number analyzed (Participants) | 100
mm | 0.23 [0.16 to 0.29]

ADVERSE EVENTS:
Time Frame: Adverse event information was collected through 12 months.
Description: The same participant may be included in more than one category therefore the number of participants does not equal the total number of participants in the group.
Arm/Group | SYNERGY Stent System
Serious Adverse Events (participants affected / at risk) | 38/100
Other Adverse Events (participants affected / at risk) | 73/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SYNERGY Stent System (N=100)
Coronary Artery Dissection (Cardiac disorders) | 7 (7)
Angina Pectoris (Cardiac disorders) | 6 (6)
Myocardial Ischemia (Cardiac disorders) | 3 (3)
Coronary Artery Stenosis (Cardiac disorders) | 2 (2)
Palpitations (Cardiac disorders) | 2 (2)
Angina Unstable (Cardiac disorders) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Presyncope (Nervous system disorders) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dizziness postrual (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Tension Headache (Nervous system disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 5 (5)
Chest discomfort (General disorders) | 1 (1)
General physical health deterioration (General disorders) | 1 (1)
Diverticulitis intestional haemorrhagic (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Meningitis (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Entropion (Eye disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Arterial rupture (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Wound drainage (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SYNERGY Stent System (N=100)
Catheter site haematoma (General disorders) | 10 (13)
Adverse drug reaction (General disorders) | 7 (8)
Non-cardiac chest pain (General disorders) | 7 (7)
Catheter site haemorrhage (General disorders) | 3 (3)
Fatigue (General disorders) | 3 (3)
Chest discomfort (General disorders) | 2 (2)
Catheter site pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 23 (23)
Angina Pectoris (Cardiac disorders) | 5 (5)
Atrial fibrillation (Cardiac disorders) | 1 (2)
Arteriospasm coronary (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Bundle branch block left (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
Headache (Nervous system disorders) | 7 (7)
Presyncope (Nervous system disorders) | 5 (7)
Syncope (Nervous system disorders) | 2 (2)
Carotid arteriosclerosis (Nervous system disorders) | 1 (1)
Dementia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dizziness ppostural (Nervous system disorders) | 1 (1)
Migrane without aura (Nervous system disorders) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 6 (6)
Back injury (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Road traffic acciedent (Injury, poisoning and procedural complications) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1)
Vascular procedure complication (Injury, poisoning and procedural complications) | 1 (1)
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1)
Helicobacter infection (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Hypotension (Vascular disorders) | 4 (4)
Arteriosclerosis (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2)
Neophrolithiasis (Renal and urinary disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1)
Blepharospasm (Eye disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Entropion (Eye disorders) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 2 (2)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Psychogenic pain disorder (Psychiatric disorders) | 1 (1)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Blood triglycerides increased (Investigations) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less